CLINICAL TRIAL: NCT02650024
Title: Impact of Hepatitis C Virus Therapy on Central Nervous System Outcomes
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ajay Bharti, Assistant Professor, University of California, San Diego
Other Study IDs: CO-US-337-1786
Record Dates: First submitted 2015-11-24; First posted 2016-01-08 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C; Human Immunodeficiency Virus
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens (including plasma EDTA and serum) are collected and batched for biomarker assays
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study observes the effects of newly developed direct-acting antiviral (DAA) treatments on the central nervous system (CNS) of individuals with chronic Hepatitis C (HCV). The goals of this study are to determine the CNS impact of curing chronic HCV disease with newly established DAA therapies and how HIV alters this relationship.

DETAILED DESCRIPTION:
The specific aims of the study are as follows:

Aim 1. Impact of HCV Cure on CNS Outcomes. Determine how curing HCV without IFN alters CNS outcomes in substance users with chronic HCV disease.

Aim 2. Correlates of CNS Outcomes. Determine the viral and host correlates of Aim 1's neurocognitive outcomes.

Aim 3. Impact of HIV Co-infection. Explore how HIV alters the relationships observed in Aims 1 and 2. Hypothesis 3: Compared with HCV mono-infected adults, SVR will be less likely to result in improved CNS outcomes in HCV/HIV co-infected adults.

ELIGIBILITY:
About 40 HCV+ and HCV/HIV co-infected patients with neurocognitive impairment (NCI) and a history of substance abuse will take part in this study.

INCLUSION CRITERIA

1. Adults (18 years old or older) with chronic HCV and NCI with a GDS greater than or equal to 0.35 (n=40).
2. Presence of chronic HCV infection based on chart review will be defined as positive for anti-HCV antibody or HCV RNA at least 6 months before screening.
3. Plan to receive HCV treatment from their primary care physician within 1 month of enrollment.
4. For the HIV/HCV co-infected group only, subjects must have HIV. HIV status will be obtained through self-report. Self-report will be confirmed at the pretreatment visit using a HIV-1 point of care test. In the event that point of care test and self-report are discordant, then HIV status will be confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV-1 and/or E/CIA, or by HIV-1 antigen, or plasma HIV-1 RNA viral load.

EXCLUSION CRITERIA

1. Cirrhosis or bridging fibrosis (mHAI stages 4-6 or its equivalent).

   * Liver biopsy at any time showing mHAI stage 4 or higher fibrosis OR
   * FibroScan within 12 months demonstrating liver stiffness of ≥9.5 kPa OR
   * APRI ≥2.0 and FIB-4 ≥3.25
   * NOTE: If APRI and FIB-4 are discordant one of the other forms of fibrosis staging must be used.
2. Any cause of liver disease other than chronic HCV infection, including but not limited to the following:

   * Hemochromatosis
   * Alpha-1 antitrypsin deficiency
   * Wilson's disease
   * Autoimmune hepatitis
   * Alcoholic liver disease
   * Drug-related liver disease
3. Severe NC confounding conditions (stroke, head injury, or developmental learning disability).
4. Regular use of anti-inflammatory drugs.
5. Current or recent treatment with pegylated interferon (PEG-IFN).
6. Other active inflammatory process (major infection, malignancy, rheumatoid arthritis/autoimmune disorder) within the prior 28 days.
7. Uncontrolled or active depression or other psychiatric disorder that in the opinion of the site investigator might preclude adherence to study requirements or impact NC functioning and assessments.
8. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
9. Presence of active or acute AIDS-defining opportunistic infections within 12 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 75% of subjects will be male and 25% female. Based on the nature of the HCV clinics where the cohort will be largely recruited, we expect to enroll approximately 25-30% Hispanics, 15-20% African Americans, 2-5% Asian-Pacific Islanders, and 50% non-Hispanic whites.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with change in neurocognitive impairment defined by Global Deficit Score (GDS) > or equal to 0.5 related to HCV treatment | 5 years
  Neurocognitive impairment, defined as GDS > or equal to 0.35, will be tested using a battery of tests covering 7 neurocognitive ability domains that include verbal fluency, information processing speed, learning, memory, executive functions, attention and working memory, fine motor skills.

SECONDARY OUTCOMES:
Number of participants with abnormal laboratory values representing viral and host factors related to HCV treatment | 5 years
  Viral factors: i) HCV RNA: will be measured according to the manufacturer's instructions (limit of detection 30 IU/mL). Enzyme-linked immunosorbent assay (ELISA) kits or multiplex assays will be used for measuring soluble biomarkers in cerebrospinal fluid (CSF) and plasma. ii) HCV core protein: Quantitative ELISA (limit of detection 1 ng/mL). Host factors: i) Neurofilament-light: Quantitative ELISA (limit of detection 50 pg/mL). ii) Soluble tumor necrosis factor receptor-II (sTNFR-II): Quantitative ELISA (limit of detection 2.3 pg/mL). iii) Macrophage Inflammatory protein--1β (MIP-1β), Interleukin-18 (IL-18) and Interferon gamma-induced protein-10 (IP-10). iv) sCD14: (sensitivity 125 pg/mL). v) sCD163: (limit of detection 0.613 ng/mL). vi) Neopterin: Quantitative ELISA (limit of detection 0.7 nmol/L).
Number of HIV-infected participants with abnormal laboratory values representing viral and host factors related to HCV treatment | 5 years
  Neurocognitive performance and viral and host biomarkers will be measured as mentioned above.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Bharti, M.D., Principal Investigator — UCSD
Locations (1):
- Ucsd Hnrp, San Diego, California, United States